CLINICAL TRIAL: NCT05534269
Title: Stress Urinary Incontinence Study to Assess Safety and Efficacy of Muvon's Muscle Precursor Cell Therapy
Acronym: SUISSE MPC2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: GCP-Service International Ltd. & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUISSE MPC2
Record Dates: First submitted 2022-08-23; First posted 2022-09-09 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Female Stress Urinary Incontinence
Keywords: SUI; Incontinence; rhabdomyosphincter; urine; Stress Incontinence; LUTS; lower urinary tract
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Low dose and High dose evaluation
Who Masked: Participant
Masking Description: Neither patient nor sponsor will know which patient gets which dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose (Experimental): Already human tested low dose from phase I study
  Interventions: Biological: autologous muscle precursor cells
- High dose (Experimental): First in human dose used for efficacy reasons during phase II
  Interventions: Biological: autologous muscle precursor cells

INTERVENTIONS:
Biological: autologous muscle precursor cells — Patients own Muscle Precursor Cells are isolated and injected into the rhabdomyosphincter

SUMMARY:
The objective of the SUISSE MPC 2 study is to treat stress urinary incontinence in adult women.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) is the loss of small amounts of urine associated with coughing, laughing, sneezing, exercising or other activities that increase pressure on the abdomen and, subsequently, the bladder.

The goal of the SUISSE MPC2 study is to treat SUI in women using their own autologous muscle precursor cells. To generate enough outcome data, a sufficient number of patients will be enrolled to yield evaluable data from 30 patients.

The study will be conducted as a self-controlled case series (SCCS) with each patient serving as their own comparators. Patients will participate in the study for up to approximately 8 to 9 months, including a baseline visit for screening, a visit to obtain a muscle biopsy approximately 12 weeks later, an injection of MPCCOLs up to 5 weeks later, and follow-up visits at 1, 3 and 6 months post injection. The injection is performed with ultrasound guidance using an endocavity ultrasound probe mounted on an Injection Device specifically designed for the clinical trial.

All patients will be treated with one of two doses of MPCCOL, assigned according to the study's randomization method.

Half of the participating patients will receive the tissue engineered product (TEP) dose that was previously studied in the completed phase I study. The other half of the participants will receive a higher dose of the cell therapy to investigate the effects of dose increase. All study participants will be monitored via medical examinations.

Separate from the Principal Investigator, safety events will be reported to and investigated by an independent Data Safety Monitoring Board (DSMB) consisting of independent physicians and experts in the field. Data regarding the functionality and safety of the Injection Device will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Predominant clinical diagnosis of SUI
* Stress incontinence ≥ grade I for at least 6 months
* Patient has at least once been treated with, and failed prior conservative treatments
* Patient had no improvement of SUI symptoms for at least 6 months before enrollment
* Patients with a certain amount of leaks or /and a predefined pad weight at screening
* Candidate for a surgical treatment
* Negative blood test: Human immunodeficiency virus (HIV 1/2), Hepatitis B HBsAg, Anti HBc, Hepatitis C, Anti-HCV-Ab and Syphilis
* Negative laboratory or blood test, and medical examination to eliminate risk of sexually transmitted diseases (STD) per investigators' discretion
* Competent to comprehend, sign, and date informed consent form before any study-specific procedure is performed
* Able to communicate well with the Investigator, and to understand and comply with the requirements of the study including answering the required questionnaires

Exclusion Criteria:

* History of anti-incontinence surgery or prolapse surgery.
* Prolapse
* Diagnosed Hypermobile Urethra
* Previous diagnosis of any of the following conditions, disorders, or diseases of the urinary tract:

  * Clinically significant cystocele or rectocele
  * Ureteric bladder, urethral or rectal fistula
  * Uncorrected congenital abnormality leading to urinary incontinence
  * Interstitial cystitis
* Urinary urgency that results in leakage (as a predominant symptom)
* Adult enuresis
* Urodynamically proven detrusor instability or detrusor sphincter dyssynergia (DSD)
* Sensory urgency defined as first sensation of bladder fill (urge to void) of <100 ml
* No sensation at any time during the simple filling cystometry procedure
* Known urethral Stenosis (ureterocystoscopy) or urethral diverticulum
* History of cancer (< 5 year of remission) or history of pelvic radiotherapy
* Immunosuppressed patients
* Women who are pregnant or become pregnant during the course of the study, breast feeding or <12 months postpartum
* Untreated symptomatic urinary tract infection
* Fever (as defined by ≥ 38,5°C, axillar measurement), any infectious disease, cold or flu within the last 7 days
* Unstable severe systemic disease including uncontrolled hypertension, unstable angina, or myocardial infarction, severe coagulation disorders, bleeding diathesis, emboli, thrombophlebitis, infectious diseases, poor wound healing, and poorly controlled diabetes mellitus within 6 months before enrolment
* Known allergy/intolerance to at least one of the active ingredients or excipients of the investigational products
* Known allergy/intolerance to Penicillin or Streptomycin.
* Known genetically determined or acquired muscular disease, known neurological disorder (Parkinson's disease, multiple sclerosis, spina bifida, medullary traumatism, Creutzfeldt-Jakob disease).
* Medication regimen including estrogens, anti-estrogens or diuretics where dose and/or frequency has not been stable for at least the past 12 weeks or is anticipated to change during the course of the study.
* Chronic use of defined drugs and not stopped prior to inclusion into or including the study. Selective serotonin and norepinephrine reuptake inhibitor antidepressant (SSNRI), alpha-receptor antagonists/agonists, beta-3-receptor agonists or anticholinergic/-muscarinic drugs.
* Have any clinically significant coexisting condition or symptoms that, in the opinion of the investigator, would put the safety of the participant at risk.
* Any organic or psychiatric disorder that, in the opinion of the investigator, might prevent the subject from completing the study or interfere with the interpretation of the study results.
* Medication known to affect lower urinary tract function.
* Patients having any electrical device inside their body (such as a cochlear implant, TENS stimulator (for pain), vagal nerve stimulator, brain stimulator, gastric pacemaker, bladder stimulator, or an implanted mechanical pump (such an insulin pump or pain pump).
* Patients having a cardiac pacemaker or defibrillator implant.
* Patients with Starr-Edwards artificial heart valve.
* Patients that suffer from claustrophobia.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Change of SUI episode frequency | 8-9 months
  Assessment in episode change measured using a bladder diary, from baseline to 6 months after injection.

SECONDARY OUTCOMES:
Incidence of (S)AEs | 6-8 months
  AEs related to obtaining biopsy, injection procedure and MPCs, including surgical injury, scars, urinary tract infection, inflammation, pelvic pain, prolonged urinary retention, voiding dysfunction, de novo urge incontinence, haematuria, aberrant tissue formation.
  Measured from Visit 2 (biopsy) to End of Study.
Number of patients with any clinical significant findings | 8-9 months
  Number of patients with any clinically significant findings based on physical examination, standard haematology, clinical chemistry and urinalysis profiles, blood pressure (BP), pulse and adverse events recordings at baseline, 1 month, 3 months and 6 months post-implantation.
Change in 24 hour pad weight | 8-9 months
  Change in pad weight based on using regular pad tests, from baseline to 6 months after injection.

OTHER OUTCOMES:
Change in total leakage episodes | 8-9 months
  Response rate at 6 months, defined as percentage of patients with at least 50% change in number of stress leaks
Questionnaire ICIQ-UI SF (International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form ) | 8-9 months
  Change in score from baseline to 6 months. Containing 1 scale ranging from 0 (not at all) to 10 (serious) measuring the impairment caused by urine leakage in everyday life.
Questionnaire ICIQLUTSqol (International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms quality of Life) | 8-9 months
  Change in score from baseline to 6 months. This questionnaire contains 21 questions to measure the impact of urinary incontinence on quality of life with particular reference to social effects. Each question is accompanied by a scale to capture the subjective restriction concerning the respective topic. These scales range from 0 (not at all) to 10 (very much).
Questionnaire VAS (Visual analogue scale) | 8-9 months
  Change score for degree of suffering, quality of life overall and subjective health status from baseline to 6 months. Scales ranging from 0 to 10. For Quality of life and health status from 0 "very bad" to 10 "very well". The degree of suffering from 0 (low) to 10 (high).
Urethral pressure profile | 8-9 months
  It measures the changes in the bladder pressure (in cm/H2O) required to urinate and the flow rate (in ml/s) a given pressure generates between baseline and 6 months after injection.
Urodynamic cystometric test | 8-9 months
  It measures the change of how much urine (in mL) the bladder can hold, between baseline and 6 months after injection.
Urodynamic cystometric test | 8-9 months
  It measures the change how much pressure builds up inside the bladder (in cm/H2O) as it stores urine, between baseline and 6 months after injection.
Urodynamic cystometric test | 8-9 months
  It measures the change how full the bladder is (in mL) when the urge to urinate occurs, between baseline and 6 months after injection.
Urodynamic leak point pressure measurement | 8-9 months
  It measures the changes of pressure (in cm/H2O) at the point of leakage between baseline and 6 months after injection.
% of subjects with successful injection | 1 day
  at day of implantation
MRI evaluation: Increase of sphincter diameter and (S)AEs | 8-9 months
  MRI examinations of the rhabdomyosphincter at baseline visit and after ca. 6 months after the MPC injection at the end of the study. This means approximately 8-9 months after the baseline visit.
  During the MRI we will measure the increase in sphincter diameter as well as looking for potential aberrant tissue formation and necrosis. The outcome will be reportet via MRI-pictures and data measurement provided by a Radiologist via the internal hospital system.
PGI-I Questionnaire | 8-9 months
  Response to Patient Global Impression of Improvement Questionnaire, ca. 6 months after MPC injection at end of study visit.
Device deficiency, ADEs and SADEs related to the Injection Device | 6-8 months
  Device deficiencies and Adverse Device Events and Serious Adverse Device Events regarding the Injection Device used during the MPC injection step.
1 hour pad test | 6-8 months
  Reduction in weight of standardized 1 hour pad test; From visit 3 (injection) to end of study visit. The pad test will be performed at the clinic under supervision of a member of the study personnel.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Schmidli, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website for Phase II Study — http://www.muvon-trials.com